CLINICAL TRIAL: NCT00933283
Title: A Phase I, Open-Label, Single-Sequence Drug-Drug Interaction Trial in Subjects on Stable Methadone Maintenance Therapy, to Investigate the Potential Interaction Between Telaprevir 750 mg q8h and Methadone, at Steady-State
Brief Title: A Study to Investigate the Potential Interaction Between Telaprevir and Methadone, at Steady-State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015931; VX-950-TiDP24-C135 (Other: Tibotec-Virco Virology BVBA)
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Participants
Keywords: Healthy participants; Pharmacokinetics; Pharmacodynamic; Potential interaction; VX-950-TiDP24-C135; VX-950; Methadone; Telaprevir; Steady-state
MeSH Terms: interventions — telaprevir; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telaprevir + Methadone (Experimental): Patients will receive telaprevir 750 mg orally, every 8 hours from Day 1 to Day 7, along with methadone 30 to 130 mg, once daily.
  Interventions: Drug: Telaprevir; Drug: Methadone

INTERVENTIONS:
Drug: Telaprevir — Telaprevir 750 mg will be administered orally, every 8 hours from Day 1 to Day 7, along with methadone, once daily.
Drug: Methadone — Methadone 30 to 130 mg will be administered as a stable oral therapy from Day -14 to Day -1, in combination with telaprevir from Day 1 to Day 7, and then alone as a continued intake dose for an additional 30 to 32 days.

SUMMARY:
The purpose of this study is to evaluate the effect of steady-state (constant concentration of medication in the blood) telaprevir 750 mg every 8 hours on the steady-state pharmacokinetics (how the drug concentrations change over time) of R- and S-methadone.

DETAILED DESCRIPTION:
This is a Phase 1, open-label (all people know the identity of the intervention), single-sequence study to evaluate the potential interaction of steady-state telaprevir on the steady-state pharmacokinetics of methadone. The study consists of 3 phases: the screening phase (within 21 days prior to the start of supervised methadone intake on Day -14), treatment phase, and follow-up phase. Participants on stable methadone maintenance therapy will be enrolled in this study and their methadone doses will not be changed starting at Day -14. During the treatment phase, telaprevir will be added for 7 days (from Day 1 to Day 7) to participants' current methadone therapy. The methadone dosage will not to be changed from Day -14 until Day 7. All the intakes of methadone and telaprevir will be supervised and pharmacokinetic parameters will be measured during the study. Safety evaluations for adverse events, clinical laboratory tests, alcohol breath test, cardiovascular safety, and other evaluations (physical examination, and pharmacodynamic assessments) will be performed throughout the study. The total duration of the study for each participant is approximately 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Must receive once daily oral methadone maintenance therapy at a stable individualized dose of 30 to 130 mg for at least 2 weeks prior to screening, formulated as commercially available tablets or solution
* Must agree not to change the current methadone dose from screening until Day 7 included to have a daily observed and documented methadone intake from Day -14 until Day 8 and a daily observed and documented telaprevir intake from Day 1 until Day 7
* Participants have to obtain approval for participation from his/her addiction physician, and the addiction physician has to agree to provide medical care for the participant after discharge from study center
* General medical condition must not interfere with the assessments and the completion of the study
* Health assessments will be done on the basis of physical examination, medical history, electrocardiogram, vital signs and the results of blood biochemistry, blood coagulation and hematology tests and a urinalysis carried out at screening

Exclusion Criteria:

* History of any illness that could confound the results of the study or pose an additional risk in administering study medication to the participant, for eg, history of relevant medication or food allergies, history of cardiovascular or central nervous system disease, history or presence of clinically significant pathology or history of mental disease
* Consumption of herbal medications or dietary supplements, vitamins, and grapefruit or grapefruit juice, apple juice or orange juice within 14 days before Day -1
* Current alcohol use, which, in the assessment of the investigator, could compromise participant's safety or compliance with the study protocol procedures
* Test positive for drugs of abuse such as cocaine, amphetamines, barbiturates, benzodiazepines, or opiates on Day -2 unless explained by allowed concomitant medications
* Participation in a clinical study involving administration of an investigational medication within 60 days or 5 half-lives (whichever was longer) prior to the screening visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of telaprevir | On Day 7
  Pharmacokinetic parameter Cmax of telaprevir is measured when telaprevir will be administered at 750 mg every 8 hours for 7 days added to stable methadone maintenance therapy.
Minimum plasma concentration (Cmin) of telaprevir | On Day 7
  Pharmacokinetic parameter Cmin of telaprevir is measured when telaprevir will be administered every 8 hours for 7 days added to stable methadone maintenance therapy.
Area under the plasma concentration-time curve (AUC) of telaprevir | On Day 7
  Pharmacokinetic parameter AUC of telaprevir is measured when telaprevir will be administered every 8 hours for 7 days added to stable methadone maintenance therapy.
Cmax of R-methadone | Day -1 and Day 7
  Pharmacokinetic parameter Cmax of R-methadone is measured during stable methadone maintenance therapy alone and in the presence of steady-state telaprevir at 750 mg every 8 hours.
Cmin of R-methadone | Day -1 and Day 7
  Pharmacokinetic parameter Cmin of R-methadone is measured during stable methadone maintenance therapy alone and in the presence of steady-state telaprevir every 8 hours.
AUC of R-methadone | Day -1 and Day 7
  Pharmacokinetic parameter AUC of R-methadone is measured during stable methadone maintenance therapy alone and in the presence of steady-state telaprevir every 8 hours.
Cmax of S-methadone | Day -1 and Day 7
  Pharmacokinetic parameter Cmax of S-methadone is measured during stable methadone maintenance therapy alone and in the presence of steady-state telaprevir at 750 mg every 8 hours.
Cmin of S-methadone | Day -1 and Day 7
  Pharmacokinetic parameter Cmin of S-methadone is measured during stable methadone maintenance therapy alone and in the presence of steady-state telaprevir every 8 hours.
AUC of S-methadone | Day -1 and Day 7
  Pharmacokinetic parameter AUC of S-methadone is measured during stable methadone maintenance therapy alone and in the presence of steady-state telaprevir every 8 hours.

SECONDARY OUTCOMES:
Short Opiate Withdrawal Scale [SOWS] | Day -7, and Day -2 to Day 7
  Pharmacodynamic assessments of methadone withdrawal are performed by means of SOWS.
Desires for Drugs Questionnaire [DDQ] | Day -7, and Day -2 to Day 7
  Pharmacodynamic assessments of methadone withdrawal are performed by means of DDQ.
Pupillometry | Day -1, Day 2, Day 4, and Day 7
  Pharmacodynamic assessments of methadone withdrawal are performed by means of pupillometry.
Number of participants with adverse events | Up to 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA

REFERENCES:
- [Derived] van Heeswijk R, Verboven P, Vandevoorde A, Vinck P, Snoeys J, Boogaerts G, De Paepe E, Van Solingen-Ristea R, Witek J, Garg V. Pharmacokinetic interaction between telaprevir and methadone. Antimicrob Agents Chemother. 2013 May;57(5):2304-9. doi: 10.1128/AAC.02262-12. Epub 2013 Mar 11. PMID 23478952
- See also: A Phase I, open-label, single-sequence drug-drug interaction trial in subjects on stable methadone maintenance therapy, to investigate the potential interaction between telaprevir 750 mg q8h and methadone, at steady-state. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1069&filename=CR015931_CSR.pdf